CLINICAL TRIAL: NCT00384956
Title: A Phase II Study of Intravenous Azacitidine Alone in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0585
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS either de novo or secondary, fitting any of the WHO classifications.
MeSH Terms: conditions — Myelodysplastic Syndromes; Neoplasm Metastasis | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine (Experimental): Azacitidine 75 mg/m2 IV on days 1-5 of each 28 day cycle. Patients that do not respond after two cycles will have the dose increased to 100 mg/m2. Patients who achieve a CR will receive 3 additional 28 day cycles and then begin treatment on days 1-5 of a 56 day cycle. Individuals who demonstrate a loss of response will resume 28 day cycles.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine
  Other Names: 5-azacitidine; Vidaza

SUMMARY:
The primary endpoint of this study is to estimate morphologic complete remission rate. Estimation of response rate is also a secondary objection.

DETAILED DESCRIPTION:
Myelodysplastic syndrome (MDS) is a hematological disorder characterized by ineffective hematopoiesis. The only known curative treatment for patients with MDS is allogeneic stem cell transplantation. However, only a minority of patients are candidates for this aggressive therapy. DNA hypomethylation agents have been shown to have activity in this disorder and are postulated to work by reversing this epigenetic mechanism of gene-silencing. Recently, 5-azacitidine, administered subcutaneously for seven days, received approval by the FDA for the therapy of MDS based on a randomized trial which demonstrated a diminished risk of leukemic transformation and improved survival when compared to best supportive care.

The subcutaneous route of administration can present challenges to implementing this therapy. In the CALGB studies 8921 and 9221, approximately 23% of patients had significant injection site pain. Moreover, 35 % of patients had injection site bruising which can be extensive in thrombocytopenic patients. Due to limitations on drug concentration and administration volumes for subcutaneous dosing, patients often need to have two or three injections at separate sites each day to meet target dosing. In addition, the schedule of administration is inconvenient in an outpatient setting secondary to the need to schedule administrations over weekends. Therefore, there is great interest in pursuing an abbreviated intravenous route for administration of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological MDS either de novo or secondary, fitting any of the FAB classifications, confirmed by institutional pathologist within 2 weeks prior to start of treatment. Patients with 5% bone marrow blasts must also meet one of the following criteria:

   * Symptomatic anemia with either hemoglobin less than 10.0 g/dL or requiring RBC transfusion
   * Thrombocytopenia with a history of two or more platelet counts < 50,000 / µL or a significant hemorrhage requiring platelet transfusions, or
   * Neutropenia with two or more absolute neutrophil counts less than 1,000 /µL.
2. ECOG performance status of 0-2.
3. Must give written informed consent indicating their awareness of the investigational nature of this study and its potential hazards.
4. Adequate renal and hepatic function (creatinine ≤ 150% of institutional upper limit of normal, total bilirubin ≤ 150% institutional upper limit of normal, AST ≤ 200% institutional upper limit of normal).
5. Life expectancy of at least 12 weeks.
6. Have not received any chemotherapy within 4 weeks of study enrollment and must have recovered from any treatment-related toxicities.
7. Women of childbearing age must have a negative serum pregnancy test prior to initiating therapy.
8. Sexually active women of childbearing potential must use effective birth control during the trial and for an appropriate period after the trial.
9. Men must be willing to avoid fathering a new child while receiving therapy with azacitidine.
10. ≥18 years, no upper age limit
11. Individuals who are candidates for hematopoietic stem cell transplantation and who meet all other study criteria may participate in the study and receive intravenous azacitidine alone as a treatment prior to transplantation.

Exclusion Criteria:

1. Known CNS leukemia.
2. Previously received Azacitidine (Vidaza®, Pharmion Corp., Boulder CO) or decitabine (Dacogen®, MGI Pharma Inc. Bloomington, MN).
3. Known or suspected hypersensitivity to azacitidine or mannitol.
4. Receiving any other investigational agents within 30 days of first dose of study drug.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure of NYHA class 3 or 4, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
6. Known positive serology for HIV.
7. Had radiotherapy within 14 days prior to study enrollment.
8. Known presence of hepatic tumors.
9. <18 years of age
10. Exclude women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study started on 08/17/2006 and enrollment to the study closed on 06/10/2008.
Period: Overall Study
Arm/Group | Azacitidine
Started | 25
Completed | 22
Not Completed | 3
Not completed — Ineligible (acute myeloid leukemia) | 3

BASELINE CHARACTERISTICS:
Population: 25 patients were enrolled and 22 were evaluable (3 patients had acute myeloid leukemia according to the FAB classification on enrollment bone marrow biopsy review and were removed from the study)
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 69.5 [53 to 79]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 22
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG Performance Status Grade
  * 0 Fully active able to carry on all predisease performance without restriction
  * 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (light house work/office work)
  * 2 Ambulatory, capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours
  * 3 Capable of limited selfcare, confined to bed/chair more than 50% of waking hours
  * 4 Completely disabled. Cannot carry on selfcare. Totally confined to bed/chair
  * 5 Dead
  participants
    0 | 4
    1 | 15
    2 | 2
    Unknown | 1
Duration of myelodysplastic syndrome (MDS) at study entry [Median (Full Range); unit: days] | 15.5 [0 to 1412]
French, American, British (FAB) classification [Number; unit: participants] — * RA = refractory anemia
  * CMML = Chronic myelomonocytic leukemia
  * RAEB = Refractory Anemia with Excess Blasts in Transmission
  * RAEB-t =Refractory Anemia with Excess Blasts in Transformation
  participants
    RA | 6
    CMML | 2
    RAEB | 12
    RAEB-t | 2
World Health Organization (WHO) classification [Number; unit: participants] — * RA = Refractory anemia
  * RCMD = Refractory cytopenia with multilineage dysplasia
  * CMML-1 = Chronic myelomonocytic leukemia type 1
  * RAEB-1 = Refractory anemia with excess blasts type 1
  * RAEB-2 = Refractory anemia with excess blasts type 2
  * AML = Acute myeloid leukemia
  participants
    RA | 3
    RCMD | 3
    CMML-1 | 2
    RAEB-1 | 3
    RAEB-2 | 9
    AML | 2
Cytogenetics [Number; unit: participants]
  Normal | 7
  Intermediate | 4
  Complex | 11
International Prognostic Scoring System (IPSS) [Number; unit: participants] — Score values:
  * Low = 0
  * INT-1 = 0.5-1.0
  * INT-2 = 1.5-2.0
  * High = greater than or equal to 2.5
  * The two lower categories can be further described as the lower risk group while the two upper categories can be further described as the higher risk group.
  * 8 questions (7 symptoms + 1 quality of life) with answers ranging from 0=not at all to 5=almost always. The lower the score the milder the symptoms are.
  participants
    Low | 1
    Int-1 | 8
    Int-2 | 7
    High | 6
Bone marrow cellularity at baseline [Median (Full Range); unit: percentage of bone marrow cellularity] | 68 [20 to 90]
Transfusion dependence [Number; unit: participants] — Only 10 out of 22 evaluable participants have baseline transfusion dependence.
  participants
    Red blood cell | 4
    Platelet | 3
    Red blood cell and platelet | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission (CR) and Partial Remission (PR)
Description: Defined according to the modified International Working Group (IWG) (2006) response criteria for myelodysplasia:
  CR=bone marrow with <5% myeloblasts and 0% peripheral blasts, hemoglobin ≥11g/dL, platelets ≥ 100 x 10^9/L, and neutrophils ≥1.0 x 10^9/L. Residual dysplasia was allowed.
  PR= All of the CR criteria if abnormal before treatment except: bone marrow blasts decreased by ≥50% over pretreatment but still >5%.
Time Frame: After 4 cycles of therapy (up to 112 days after start of treatment)
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
participants
  Complete remission (CR) | 5
  Partial remission (PR) | 1

2. Secondary Outcome: Rate of Hematologic Improvement
Description: International Working Group (IWG) for Myelodysplasia (MDS).
Time Frame: 4 weeks following last azacitidine dose [median number of cycles 4.5 (1-20)]
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
participants | 0

3. Secondary Outcome: Rate of Transfusion Independence
Time Frame: 4 weeks following last azacitidine dose [median number of cycles 4.5 (1-20)]
Population: Only participants with baseline transfusion dependence were assessed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 10
participants
  Red blood cell | 2
  Platelet | 1
  Red blood cell and platelet | 0

4. Post Hoc Outcome: Time to Best Response
Time Frame: 4 weeks following last dose of azacitidine [median number of cycles 4.5 (1-20)]
Measure: Median (Full Range); unit: days
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
days | 108 [27 to 192]

5. Secondary Outcome: Rate of Cytogenetic Response
Time Frame: 2 years after first dose of study drug or until participant is lost to follow-up or dies
Population: This secondary outcome was not analyzed.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Overall Survival
Description: Overall survival is defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: 2 years after first dose of study drug or until participant is lost to follow-up or dies
Measure: Median (Full Range); unit: days
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
days | 444 [23 to NA] — At the time the data was analyzed, the upper range of overall survival was not reached.

7. Secondary Outcome: Rate of Relapse After Hematopoietic Stem Cell Transplant in Individuals Treated With 5-azacitidine Prior to Transplant.
Time Frame: 2 years after first dose of study drug or until participant is lost to follow-up or dies
Population: This secondary outcome was not analyzed.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Duration of Response (DOR)
Time Frame: 2 years after first dose of study drug or until participant is lost to follow-up or dies
Measure: Median (Full Range); unit: days
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
days | 450 [169 to NA] — At the time that the data was analyzed, the upper range for DOR had not been reached.

9. Post Hoc Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause.
  Disease progression
  * for patients w/ <5% blasts; a ≥50% increase in blasts to >5% blasts
  * for patients w/ 5% to 10% blasts; a ≥50 increase to >10% blasts
  * for patients w/ 10% to 20% blasts; a ≥50% increase to >20% blasts
  * for patients w/ 20% to 30% blasts; a ≥50% increase to >30% blasts
  * One or more of the following ≥50% decrement from maximum remission/response levels in granulocytes or platelets, reduction in hemoglobin concentration by ≥2 g/dL or transfusion dependence
Time Frame: 2 years after first dose of study drug or until participant is lost to follow-up or dies
Measure: Median (Full Range); unit: days
Arm/Group | Azacitidine
Number analyzed (Participants) | 22
days | 339 [32 to NA] — At the time the data was analyzed, the upper range of PFS was not reached.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 4 weeks following last dose of azacitidine.
Description: 24 patients out of 25 patients received at least the first dose of azacitidine. One patient was enrolled in the study but did not receive treatment due to a catheter port infection.
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 12/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=24)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with unknown neutrophils (sepsis) (Infections and infestations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Infection (sepsis) (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
Chills (General disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Neutropenic fever (Infections and infestations) | 5
Death due to progressive disease (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Infection without neutropenia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=24)
Abdominal pain (Gastrointestinal disorders) | 3
Alkaline phosphatase (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bilateral lower extremity edema (General disorders) | 5
Bilateral upper extremity edema (General disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 4
Chest/ribs pain (Musculoskeletal and connective tissue disorders) | 5
Colitis (Gastrointestinal disorders) | 3
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 6
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Elevated creatinine (Investigations) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Face pain (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 8
Fever - no infection (General disorders) | 4
Headache (Nervous system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 14
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Hyperbilirubinemia (Investigations) | 8
Hypercalcemia (Investigations) | 2
Hyperglycemia (Investigations) | 9
Hyperkalemia (Investigations) | 5
Hypermagnesemia (Investigations) | 4
Hypernatremia (Investigations) | 4
Hypertension (Cardiac disorders) | 1
Hypoalbuminemia (Investigations) | 11
Hypocalcemia (Investigations) | 9
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 5
Hyponatremia (Investigations) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Infection with neutropenia (Infections and infestations) | 9
Insomnia (Psychiatric disorders) | 2
Left apical mass (General disorders) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 2
Lesion (Skin and subcutaneous tissue disorders) | 1
Leukocytes (WBC) (Investigations) | 11
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Investigations) | 4
Mental status change (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 1
Mucositis (Gastrointestinal disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal drainage/congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Neutropenic fever (Infections and infestations) | 1
Neutrophils (ANC) (Investigations) | 13
Oral cavity hemorrhage (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Petechiae (Blood and lymphatic system disorders) | 2
Platelets (Investigations) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Right abdominal infection (Gastrointestinal disorders) | 1
Right lower quadrant mass (General disorders) | 1
Rigors/chills (General disorders) | 4
SGOT (AST) (Investigations) | 7
SGPT (ALT) (Investigations) | 9
Sensory neuropathy (Nervous system disorders) | 2
Somnolence (Psychiatric disorders) | 1
Subclavian nodularity (General disorders) | 1
Sweating (General disorders) | 1
Tachycardia (Cardiac disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Upper extremity pain (Musculoskeletal and connective tissue disorders) | 2
Uric acid (Investigations) | 3
Urinary urgency (Renal and urinary disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes